CLINICAL TRIAL: NCT06186258
Title: Infective Endocarditis in Percutaneous Pulmonary Revalvulation: a Direct Comparison Between Melody and Sapien Valves
Brief Title: Infective Endocarditis in Percutaneous Pulmonary Revalvulation: Comparison Between Melody and Sapien Valves
Acronym: Endopulm
Status: Completed | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-552
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Infective Endocarditis; Congenital Heart Disease; Percutaneous Pulmonary Valve Implantation
Keywords: percutaneous pulmonary valve implantation; Sapien 3; Melody; Transcatheter pulmonary valve replacement; infective endocarditis; congenital heart disease
MeSH Terms: conditions — Endocarditis; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Patients who underwent successful percutaneous pulmonary revalvulation with the Melody valve: Data from patients managed for a pulmonary revalvulation procedure with the Melody valve between 01/01/2007 and 31/12/2021 will be collected.
  Cases of infective endocarditis will be meticulously examined and classified as certain, possible or refuted, according to the modified Duke algorithm proposed by the European Society of Cardiology.
  Cases of endocarditis occurring within one year of pulmonary revalvulation will be classified as early IE and other cases as late IE
  Interventions: Device: percutaneous pulmonary valve implantation (PPVI)
- Patients who underwent successful percutaneous pulmonary revalvulation with the Sapien 3, XT valve: Data from patients managed for a pulmonary revalvulation procedure with the Sapien 3, XT valve between 01/01/2007 and 31/12/2021 will be collected.
  Cases of infective endocarditis will be meticulously examined and classified as certain, possible or refuted, according to the modified Duke algorithm proposed by the European Society of Cardiology.
  Cases of endocarditis occurring within one year of pulmonary revalvulation will be classified as early IE and other cases as late IE
  Interventions: Device: percutaneous pulmonary valve implantation (PPVI)

INTERVENTIONS:
Device: percutaneous pulmonary valve implantation (PPVI) — The only inclusion criterion is a successful PPVI to treat RVOT dysfunction. Procedural techniques were at each operator's discretion as well as post-procedure treatments and patient's follow-up. As we sought to assess IE incidence during follow-up, patients who underwent catheterization for intended PPVI but who did not had a successful valve implantation were not included. Successful PPVI was defined as patient discharged alive without valve surgery after successful valve implantation in the RVOT.

SUMMARY:
Percutaneous pulmonary valve revalvulation (PPVR) has emerged as an alternative to surgery for the treatment of congenital heart disease with right ejection pathway dysfunction. The Melody valve (Medtronic Inc., Minneapolis, Minnesota) was the first to be used, validated in 2006 by the European Commission and in 2010 by the Food and Drug Administration (FDA). Subsequently, the Sapien valve (Edwards SAPIEN pulmonic transcatheter heart valve, Edwards Lifesciences, Irvine, California) was subsequently approved for PPVR (Europe, 2010; FDA 2016).

Infective endocarditis (IE) after PPVR is currently a major concern with an incidence after Melody PPVR estimated at 3%, much higher than the rate of prosthetic left-heart IE. The Sapien valve has been introduced more recently and some cases of IE have been published. Despite the attention this issue is receiving, there are few studies of sufficient size or statistical power to elucidate the risk factors for developing an IE after PPVR according to the type of valve implanted. Recently, a multicenter study was published by the American team of McElhinney et al (J Am Coll Cardiol 2021 ; 78 :575-589). Although it was a sizeable cohort (2476 patients), there was a large disparity in the ratio of patients who underwent revalvulation with either the Melody or Sapien valve, in favor of Melody patients (2038 Melody patients vs. 438 Sapien patients). In this study, the estimated risk of IE was higher for patients who received a Melody valve, according to univariable analysis but not anymore after multivariate analysis. To further answer this question, we develop an international retrospective multicenter registry whose main objective will be to characterize the incidence rate of infective endocarditis after percutaneous pulmonary revalvulation according to the type of valve implanted (Melody vs. Sapien) using a large population of patients with comparable characteristics (match-population).

DETAILED DESCRIPTION:
Infective endocarditis (IE) is a dreaded complication in patients with congenital heart disease (CHD), with an incidence up to 100-fold compared to the general population. In CHD such as cono-truncal defects, the right ventricular outflow tract (RVOT) is reconstructed using patches, conduits, homografts or bioprosthetic valves. Subsequently, pulmonary regurgitation, conduit degeneration, or conduit mismatch due to growth may require repeated valve and/or conduit replacement. Transcatheter pulmonary valve implantation (TPVI) is an effective treatment for RVOT dysfunction, as an alternative to surgical pulmonary valve replacement. TPVI was first described in 2000 and, since then, many studies have supported its safety and efficacy. The MELODY valve (Medtronic Inc., Minneapolis, MN) was used first and received European certification in 2006 and FDA approval in 2010. The SAPIEN valve series (Edwards SAPIEN pulmonic transcatheter heart valve, and SAPIEN 3 valve, Edwards Lifesciences, Irvine, CA) were subsequently licensed for TPVI (Europe 2010; and FDA, 2016). The feasibility of TPVI was initially demonstrated in right ventricle-to-pulmonary artery conduits and then in bioprostheses, small expandable conduits, and native or patched RVOTs. IE after TPVI (TPVI-IE) remains a life-threatening adverse event that affects valve durability and patient outcomes. National and international recommendations provide only meager guidance about the management of TPVI-IE. A history of IE, Di George syndrome, male sex, younger age at implant and increased valve gradient have been identified as risk factors for IE. However it remains a matter of debate whether the type of valve influences the risk of IE. Although the bovine jugular vein valves like the MELODY valve and the CONTEGRA conduit are mentioned as specific risk factors for IE in the German guidelines for IE, other authors did not support this in a large multicentre study. An important limitation is that most of studies had limited duration of follow-up, particularly after SAPIEN-TPVI, whereas endocarditis has been equally described many years following TPVI. The objective of this study was to identify additional risk factors for TPVI-IE over the long-term.

METHODS A retrospective study of the multicentre international ENDOCPULM registry including consecutive patients after successful MELODY and SAPIEN-TPVI between 2007 and 2021 in 35 tertiary European and Middle-East centres was designed. The study was approved by an independent ethics committee (GERM IRB 00012157, #552, December 17th, 2021) and was performed in accordance with the Declaration of Helsinki and its amendments. This report complies with STROBE guidelines for cohort studies.

ELIGIBILITY:
Inclusion Criteria:

* Minor or adult patients who have undergone a successful percutaneous pulmonary revalvulation procedure
* Patients or legal guardians who do not object to the use of their data for this research.

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient or legal guardian objecting to the use of his or her data for this research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohort will be made up of patients who have undergone successful percutaneous pulmonary revalvulation with the Melody valve, matched with patients who have undergone revalvulation with the Sapien valve (Sapien 3 and XT) between the years 2007 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
compare the risk of long-term infective endocarditis after percutaneous pulmonary revalvulation with Melody, Sapien XT, Sapien S3 valves. | 10 years
  risk of long-term infective endocarditis after percutaneous pulmonary as defined by annualized incidence of infective endocarditis

SECONDARY OUTCOMES:
Major cardiovascular events | 10 years
  MAE are defined as during follow-up: need for further surgical or percutaneous pulmonary revalvulation, transplantation, thrombosis of implanted pulmonary valve and death

CONTACTS AND LOCATIONS:
Overall Officials: Alain Fraisse, MD, PhD, Study Director — Royal Brompton & Harefield NHS Foundation Trust
Locations (18):
- France (8):
  - CHU Bordeaux, Bordeaux
  - CHU de Grenoble, Grenoble
  - Hopital Marie Lannelongue, Le Plessis-Robinson
  - CHRU Lille, Lille
  - CHU de la Timone, Marseille
  - CHU de Nantes, Nantes
  - Clinique Pasteur, Toulouse
  - CHU Toulouse, Toulouse
- Medical Hospital of the university of Munich, Munich, Germany
- Bambin Gesù Hospital,, Rome, Italy
- Hospital de Santa Marta, Centro Hospitalar Lisboa Central-EPE, Lisbon, Portugal
- King Faisal Hospital, Jeddah, Saudi Arabia
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - 12 de Octubre University Hospital,, Madrid
  - H. Ramón y Cajal University Hospital, Madrid
- United Kingdom (3):
  - Cardiology university Hospitals Birmingham, Birmingham
  - Bristol Heart Institute, University Hospitals Bristol & Weston NHS Foundation Trust, Bristol
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godart F, Baruteau AE, Petit J, Riou JY, Sassolas F, Lusson JR, Fraisse A, Boudjemline Y. Transcatheter tricuspid valve implantation: a multicentre French study. Arch Cardiovasc Dis. 2014 Nov;107(11):583-91. doi: 10.1016/j.acvd.2014.07.051. Epub 2014 Oct 2. PMID 25282331
- [Background] Hascoet S, Acar P, Boudjemline Y. Transcatheter pulmonary valvulation: current indications and available devices. Arch Cardiovasc Dis. 2014 Nov;107(11):625-34. doi: 10.1016/j.acvd.2014.07.048. Epub 2014 Oct 31. PMID 25444020
- [Background] Malekzadeh-Milani S, Houeijeh A, Jalal Z, Hascoet S, Bakloul M, Aldebert P, Piechaud JF, Heitz F, Bouvaist H, Dauphin C, Guerin P, Villemain O, Petit J, Godart F, Thambo JB, Boudjemline Y; French working group of Cardiac Catheterization in Congenital Heart Disease Patients. French national survey on infective endocarditis and the Melody valve in percutaneous pulmonary valve implantation. Arch Cardiovasc Dis. 2018 Aug-Sep;111(8-9):497-506. doi: 10.1016/j.acvd.2017.10.007. Epub 2018 Mar 9. PMID 29530718
- [Background] Hascoet S, Karsenty C, Tortigue M, Watkins AC, Riou JY, Boet A, Tahhan N, Fabre D, Haulon S, Brenot P, Petit J. A modified procedure for percutaneous pulmonary valve implantation of the Edwards SAPIEN 3 valve. EuroIntervention. 2019 Jan 20;14(13):1386-1388. doi: 10.4244/EIJ-D-18-00530. No abstract available. PMID 30327285
- [Background] Shahanavaz S, Zahn EM, Levi DS, Aboulhousn JA, Hascoet S, Qureshi AM, Porras D, Morgan GJ, Bauser Heaton H, Martin MH, Keeshan B, Asnes JD, Kenny D, Ringewald JM, Zablah JE, Ivy M, Morray BH, Torres AJ, Berman DP, Gillespie MJ, Chaszczewski K, Zampi JD, Walsh KP, Julien P, Goldstein BH, Sathanandam SK, Karsenty C, Balzer DT, McElhinney DB. Transcatheter Pulmonary Valve Replacement With the Sapien Prosthesis. J Am Coll Cardiol. 2020 Dec 15;76(24):2847-2858. doi: 10.1016/j.jacc.2020.10.041. PMID 33303074
- [Background] Le Ruz R, Plessis J, Houeijeh A, Baruteau AE, Le Gloan L, Warin Fresse K, Karsenty C, Petit J, Godart F, Hascoet S, Guerin P. Edwards SAPIEN XT transcatheter pulmonary valve implantation: 5-year follow-up in a French Registry. Catheter Cardiovasc Interv. 2021 Nov 1;98(5):990-999. doi: 10.1002/ccd.29862. Epub 2021 Jul 6. PMID 34227735